CLINICAL TRIAL: NCT02394262
Title: Prediction of Atherosclerotic Plaque Burden Progression With Sequential Coronary CT-angiography and Biomarkers
Brief Title: Sequential Coronary CT-angiography and Biomarkers
Acronym: PARSEC-NET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL49261.068.14
Record Dates: First submitted 2015-03-04; First posted 2015-03-20 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Biological Markers; Multidetector Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Serial CCTA and atherothrombosis markers (Experimental): Sequential coronary CT-angiography and assesment of biomarkers involved in atherothrombosis after 1 year follow-up.
  Interventions: Radiation: Coronary CT-angiography; Other: Assesment of biomarkers involved in atherothrombosis

INTERVENTIONS:
Radiation: Coronary CT-angiography — Sequential CCTA after one year follow-up. The first CCTA will be performed in terms of diagnostic work-up (referral outpatient Cardiology department).
Other: Assesment of biomarkers involved in atherothrombosis — Sequential assesment of atherothrombis biomarkers: baseline and at 1 year follow-up.

SUMMARY:
Currently, cardiac computed tomography angiography (CCTA) is a well-implemented non-invasive diagnostic imaging modality in patients with stable chest pain. Besides conventional CT-reading, CCTA is also capable to identify several morphologic and geometric characteristics of atherosclerotic plaques. Recently, the investigators showed that the use of semi-automated plaque quantification algorithm identified parameters predictive for acute coronary syndrome on top of clinical risk profiling and conventional CT-reading. In addition, several atherotrombosis biomarkers, like high-sensitivity cardiac troponins, are described as related to coronary artery disease and cardiovascular events. Prospective data with sequential analysis of atherosclerotic plaques combined with different atherothrombosis biomarkers are currently lacking, but will provide important clues about the pathophysiology of plaque progression and atherothrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recent history of (a)typical chest pain, who underwent a coronary calcium score scan as well as CCTA.
* Age older than 18 years and competent to perform written informed consent.
* At least 2 coronary segments with plaques:
* 1 proximal lesion.
* At least one coronary plaque consisting of a non-calcified or mixed component.

Exclusion Criteria:

* Unstable angina.
* Renal insufficiency: calculated estimated glomerular filtration rate <45mL/min.
* Iodine allergy.
* Pregnancy.
* Known history of atrial fibrillation.
* Inconclusive baseline computed coronary CT-angiography.
* Patients which are currently on oral vitamin K antagonists.
* Patients which are currently using selective anticoagulants.
* Previous PCI.
* Previous or planned coronary artery bypass grafting.
* Patients whereby the baseline CCTA was performed by a retrospective ECG-gated 'helical' protocol due to a high (>90bpm) or irregular heart rate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Plaque progression as defined by sequential CCTA using dedicated software. | 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Bas Kietselaer, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands